CLINICAL TRIAL: NCT06944847
Title: A Laboratory Study of Behavior and Performance Among People Who Vape Nicotine and/or Smoke Cigarettes - Schizophrenia Supplement
Brief Title: Vaping and Smoking Project in People With Schizophrenia
Acronym: VASP-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Roswell Park Cancer Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Larry Hawk, Ph.D., Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006122-Supplement; 3R01DA054276-03S1 (NIH)
Record Dates: First submitted 2025-04-06; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Acute Abstinence From Cigarettes vs E-cigarettes (ENDS)
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: All participants will complete two visits, one following 24-hour abstinence, the other while smoking/vaping as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily use of ENDS (Other): Participants who use nicotine-containing ENDS daily or near-daily but who do NOT smoke combustible cigarettes daily or near-daily.
  Interventions: Behavioral: Acute (24-hour) abstinence; Behavioral: Ad libitum smoking/vaping
- Daily use of combustible cigarettes (Other): Participants who smoke combustible cigarettes daily or near-daily but do NOT use nicotine-containing ENDS daily or near-daily.
  Interventions: Behavioral: Acute (24-hour) abstinence; Behavioral: Ad libitum smoking/vaping

INTERVENTIONS:
Behavioral: Acute (24-hour) abstinence — Participants will be asked to abstain from all tobacco/nicotine for 24 hours prior to the visit
Behavioral: Ad libitum smoking/vaping — Participants will be asked to smoke/vape as usual during the 24 hours prior to the visit

SUMMARY:
The proposed research will characterize withdrawal among people with schizophrenia who vape daily compared to people with schizophrenia who smoke combustible cigarettes daily, filling critical gaps in the understanding of electronic nicotine delivery systems (ENDS) dependence and contributing to the development of vaping cessation interventions amongst people with schizophrenia, the leading preventable cause of death in the US.

DETAILED DESCRIPTION:
Although withdrawal is considered a key feature of nicotine/tobacco addiction that contributes to difficulty quitting smoking and likely electronic nicotine delivery systems (ENDS; e.g., electronic cigarettes), there is currently no research on ENDS withdrawal in people with schizophrenia. The proposed supplement will conduct a systematic and comprehensive characterization of withdrawal in a sample of people with SCZ who vape daily compared to those who smoke daily, filling gaps in our understanding of ENDS dependence/withdrawal for people with SCZ and contributing to the identification of intervention targets for ENDS use.

ELIGIBILITY:
Inclusion Criteria:

* 6+ months of daily/near-daily nicotine vaping or cigarette smoking
* 200+ ng/mL cotinine on a commercially-available quick screen
* stable antipsychotic medication dose (no changes in past 6 months).

Current Exclusion Criteria:

* intention to quit daily/near-daily vaping/smoking in the next month
* current (2+ days out of the past 7) use of pipe tobacco, hookah/shisha, smokeless tobacco, dissolvable tobacco, nicotine pouches. For vaping group only, current (2+ days out of past 7) use of cigars, cigarillos, or filtered cigars that are filled with tobacco or a mix of tobacco and marijuana
* current use of any smoking cessation medication
* current severe substance dependence other than tobacco/nicotine (including cannabis; NIDA Modified ASSIST of 27+)
* current (past 2 weeks) suicidal ideation with intent and/or plan
* pregnancy (intake urine screen)
* florid psychosis or severe cognitive symptoms (score of ≥5 on PANSS items delusions (P1), hallucinatory behavior (P3), or unusual thought content (G9), conceptual disorganization (P2), abstract thinking (N5), or poor attention (G11) or a score ≥6 on grandiosity (P5) or suspiciousness (P6)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Wisconsin Smoking Withdrawal Scale - anger 0.5 | 0.5 hours
  anger subscale score
Wisconsin Smoking Withdrawal Scale - anger 2.5 | 2.5 hours
  anger subscale scores
Wisconsin Smoking Withdrawal Scale - anxiety 0.5 | 0.5 hours
  anxiety subscale scores
Wisconsin Smoking Withdrawal Scale - anxiety 2.5 | 2.5 hours
  anxiety subscale scores
Wisconsin Smoking Withdrawal Scale - sad 0.5 | 0.5 hours
  sadness subscale scores
Wisconsin Smoking Withdrawal Scale - sad 2.5 | 2.5 hours
  sadness subscale scores
Wisconsin Smoking Withdrawal Scale - conc 0.5 | 0.5 hours
  difficulty concentrating subscale scores
Wisconsin Smoking Withdrawal Scale - conc 2.5 | 2.5 hours
  difficulty concentrating subscale scores
Wisconsin Smoking Withdrawal Scale - sleep 0.5 | 0.5 hours
  sleep subscale scores
Wisconsin Smoking Withdrawal Scale - sleep 2.5 | 2.5 hours
  sleep subscale scores
Wisconsin Smoking Withdrawal Scale - appetite 0.5 | 0.5 hours
  appetite subscale scores
Wisconsin Smoking Withdrawal Scale - appetite 2.5 | 2.5 hours
  appetite subscale scores
Mood and Physical Symptoms Scale 0.5 | 0.5 hours
  single-item indicators of withdrawal facets
Mood and Physical Symptoms Scale 2.5 | 2.5 hours
  single-item indicators of withdrawal facets
Minnesota Nicotine Withdrawal Scale 0.5 | 0.5 hours
  single-item indicators of withdrawal facets
Minnesota Nicotine Withdrawal Scale 2.5 | 2.5 hours
  single-item indicators of withdrawal facets
Positive and Negative Affect Scale NA 0.5 | 0.5 hours
  negative affect subscale score
Positive and Negative Affect Scale PA 2.5 | 2.5 hours
  positive affect subscale score
Positive and Negative Affect Scale PA 0.5 | 0.5 hours
  positive affect subscale score
Positive and Negative Affect Scale NA 2.5 | 2.5 hours
  negative affect subscale score
Snaith-Hamilton Pleasure Scale 0.5 | 0.5
  Total score
Snaith-Hamilton Pleasure Scale 2.5 | 2.5 hours
  Total score
Questionnaire on Vaping Craving 0.5 | 0.5 hours
  total craving score
Questionnaire on Vaping Craving 2.5 | 2.5 hours
  total craving score
Questionnaire on Smoking Urges - Brief 0.5 | 0.5
  total craving score
Questionnaire on Smoking Urges - Brief 2.5 | 2.5
  total craving score
PhenX Toolkit Insomnia Severity Index 0.5 | 0.5
  7-item scale, with coverage of perceived impairment and interference with daily functioning
PhenX Toolkit Insomnia Severity Index 2.5 | 2.5 hours
  7-item scale, with coverage of perceived impairment and interference with daily functioning
Restlessness ratings 0.5 | 0.5
  3-item scale
Restlessness ratings 2.5 | 2.5 hours
  3-item scale
Restlessness and Agitation Questionnaire 2.5 | 2.5 hours
  11-item self-report scale total of behavioral indicators (supplemental evaluation of observer ratings)
Restlessness and Agitation Questionnaire 0.5 | 0.5 hours
  11-item self-report scale total of behavioral indicators (supplemental evaluation of observer ratings)
Identical Pairs Continuous Performance Task | Lab visits: ~2 hours
  Sustained attention, or vigilance, is the ability to maintain alertness to detect infrequent target stimuli during a long, monotonous task (e.g., Mackworth, 1948). We will use a version of the identical-pairs continuous performance task (Cornblatt et al., 1988) in which participants attend to a series of 800 4-digit numbers on a computer monitor (100-ms stimulus duration; 1500-ms ISI). Participants are asked to press the keyboard space bar only when the stimulus is identical to the immediately preceding stimulus (10% targets; Cooper et al., 2020; Rhodes & Hawk, 2016). Percent correct hits (target detections) is the primary outcome.
n-back working memory task | Lab visit ~ 2hours
  The n-back task (Strand et al., 2012; Rhodes & Hawk, 2016) requires indicating whether each stimulus in a rapidly presented series matches the location of the stimulus presented n stimuli before (n=0,1,2). Stimuli are small grey circles (100 ms; 30% targets). The focus here is on conditions that place marked demands on the "central executive" by requiring ongoing mental manipulation (i.e., n=2; see Baddeley, 2003). Brief practice with a 1- back will be followed by 2 100-trial blocks of the 2- back. Accuracy is the primary outcome.
Stop signal reaction time task | Lab visits: ~2 hours
  We will employ the stop-signal paradigm (Logan et al., 1984), which provides a relatively pure index response inhibition (e.g., Nigg, 2001). In our typical task (e.g., Hawk et al., 2018; Rhodes & Hawk, 2016), participants button press to indicate whether the "go" signal (<-- or -->) is pointing left or right. After a brief "go" practice, the stop signal (100-ms tone) is introduced, and participants complete 3 64-trail bocks during with they are asked to respond as quickly as possible but to not respond on stop signal trials (25% of trials). The stop signal occurs after go signal onset and adjusts dynamically across trials to yield
  ~50% inhibition (Logan et al., 1997). The primary outcome is stop signal reaction time (SSRT), an estimate of the speed of inhibition.
Spatial Delayed Response Task | 2 hours
  The SDR is a brief delayed-response spatial working memory task in which the participant is presented with a series of 3 screens on each trial. Screen 1 presents a dot (target stimulus) presented for at 1 of 16 locations on the computer screen. Screen 2 presents a "distractor task" that entails a sham attention task, appearing for variable 5 or 30 second delay. The distractor task involves a series of shapes presented on the screen and participants are asked to click the spacebar on the keyboard when they see a diamond, until the delay is finished. Screen 3 prompts the subject to identify the location of the target stimulus presented on Screen 1 using the mouse. Participants are prompted to respond as fast as possible, the task does not progress until the location response is recorded. Note that because the SDR was previously not sensitive to nicotine abstinence in non-psychiatric controls (Sacco, et al., 2005), we will only assess SDR changes
kcal consumed | 3 hours
  Fat, protein, and carbohydrate calories consumed
Hypothetical Commodity Purchase Tasks vaping intensity 0.5 | 0.5 hours
  intensity of demand
Hypothetical Commodity Purchase Tasks vaping intensity 2.5 | 2.5 hours
  intensity of demand
Hypothetical Commodity Purchase Tasks vaping persistence 0.5 | 0.5 hours
  persistence of demand
Hypothetical Commodity Purchase Tasks vaping persistence 2.5 | 2.5 hours
  persistence of demand
Hypothetical Commodity Purchase Tasks smoking intensity 0.5 | 0.5 hours
  intensity of demand
Hypothetical Commodity Purchase Tasks smoking intensity 2.5 | 2.5 hours
  intensity of demand
Hypothetical Commodity Purchase Tasks smoking persistence 0.5 | 0.5 hours
  persistence of demand
Hypothetical Commodity Purchase Tasks smoking persistence 2.5 | 2.5 hours
  persistence of demand
Positive and Negative Syndrome Scale positive 3 | 3 hours
  positive syndrome subscale
Positive and Negative Syndrome Scale negative 3 | 3 hours
  negative syndrome subscale
Positive and Negative Syndrome Scale general 3 | 3 hours
  general syndrome subscale

SECONDARY OUTCOMES:
modified Cigarette evaluation questionnaire | 3.5 hours
  Subjective/sensory effects of smoking expectancies will be assessed with widely used smoking measures (the modified Cigarette Evaluation Questionnaire, the short form of the Smoking Consequences Questionnaire, and the Smoking Abstinence Questionnaire) and adaptations and extensions of these measures for vaping.
modified e-Cigarette evaluation questionnaire | 3.5 hours
  Subjective/sensory effects of vaping expectancies will be assessed with widely used smoking measures (the modified Cigarette Evaluation Questionnaire, the short form of the Smoking Consequences Questionnaire, and the Smoking Abstinence Questionnaire) and adaptations and extensions of these measures for vaping.
Somatic / side effect checklist 0.5 | 0.5 hours
  Assesses a range of somatic symptoms (e.g., headaches, fatigue)
Somatic / side effect checklist 2.5 | 2.5 hours
  Assesses a range of somatic symptoms (e.g., headaches, fatigue)
Heart rate 30 | 30 minutes
  Heart rate, in beats per minute
Heart rate 60 | 60 minutes
  Heart rate, in beats per minute
Heart rate 90 | 90 minutes
  Heart rate, in beats per minute
Heart rate 120 | 120 minutes
  Heart rate, in beats per minute
Heart rate 150 | 150 minutes
  Heart rate, in beats per minute
Heart rate 180 | 180 minutes
  Heart rate, in beats per minute

OTHER OUTCOMES:
Cotinine | 0.25 hours
  assay cotinine from urine sample collected at the start of each visit in order to assess the degree of compliance with the abstinence manipulation
Expired-air carbon monoxide | 0.25 hours
  biochemical measure related to past 24-hour smoking

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hawk, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the full de-identified data set with metadata available through the National Addiction and HIV Data Archive Program (NAHDAP).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared at approximately the same time as the acceptance for publication of the main findings from the final dataset. The dataset will have a permanent digital object identifier and will be available as long as the NAHDAP is available.
Access Criteria: Per NAHDAP